CLINICAL TRIAL: NCT04084886
Title: Transcription Factor 7 Like 2 Gene Polymorphism and Advanced Glycation End Products as Risk Factors for Diabetic Nephropathy
Brief Title: TCF7L2 Gene Polymorphism and AGEs in Diabetic Nephropathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghadeer abdelrazzak mohammed, Assistant lecturer, Assiut University
Other Study IDs: TCF7L2 in Diabetic nephropathy
Record Dates: First submitted 2019-09-03; First posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Diabetic Nephropathies
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. To study genotypic distribution of the TCF7L2 gene polymorphism in Diabetic nephropathy.
2. To assess level of AGEs and Insulin in patients with Diabetic nephropathy.
3. To study correlation between polymorphism of the TCF7L2 gene, AGEs, Insulin and clinical characteristics in patients with diabetic nephropathy

DETAILED DESCRIPTION:
Diabetic nephropathy is one of microvascular complications of diabetes mellitus. DN is a multifactorial disorder that occurs in one third of patients with long standing DM. DN is one of the most serious complications that being a major contributing factor to end-stage renal disease and death in diabetic patients. The earliest clinical indication of DN is the appearance of microalbuminuria. Detection of diabetic nephropathy as early as possible, is the best chance of delaying progression to ESRD. Thus, screening for microalbuminuria is recommended annually immediately after a diagnosis of diabetes. Transcription factor 7-like 2 is a highly variable transcription factor, which is a key component of the Wnt-signaling pathway and plays a role in the regulation of insulin secretion by pancreatic beta cells and the maintenance of glucose homeostasis. TCF7L2 rs7903146 polymorphism is more associated with T2DM which mediated by decreased insulin secretion associated with defects in insulin processing, reduced effects of glucagon-like peptide-1, increased hepatic glucose production and insulin resistance. The mutant TT genotype and the T allele frequency was associated with diabetic patients who developed nephropathy. Advanced glycation end products are generated by the non-enzymatic reaction of amino groups in DNA and proteins with reducing sugars. AGEs accumulate in glomerular basement membrane. The AGEs-RAGE interaction is a causative factor for DN through activating a series of intracellular signal-cascade pathways which induce the generation of further signalling factors, such as vascular endothelial growth factor, transforming growth factor B, nuclear factor-κβ. Those signalling factors cause mesangial expansion and glomerulosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* diabetic nephropathy
* clinical diagnosis of prediabetes
* Type 2 diabetic patients

Exclusion Criteria:

* cardiovascular disease
* diabetic neuropathy
* diabetic retinopathy

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * 60 diabetic patients: Diagnosis of DM was based on the American Diabetes Association Criteria:
    -The diabetic patients will be classified into 2 subgroups:
  * 30 Diabetic patients without any microvascular or macrovascular complications.
  * 30 Diabetic patients with pure nephropathy not having other microvascular or macrovascular complications.
  * 20 patients diagnosed as prediabetes:
  * Beside 20 Apparent healthy subjects as control group.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
value of the odds ratio associated with the relationship between a polymorphism TCF7L2 gene and the occurrence of diabetic nephropathy | one year
  find a link between genetic polymorphism of TCF7L2 and the risk of developing nephropathy in diabetic patients.
  Nephropathy is defined Albumin/creatinine ratio > 30 mg/gm creat.
Number of patients with genotype TCF7L2 by PCR | 5 years
  the prevalence of TCF7L2, in the diabetic patient, and compared to the values found in the general population.
  the TCF7L2 genes will be evaluated by PCR-RFLP

REFERENCES:
- [Background] Gawandi S, Gangawane S, Chakrabarti A, Kedare S, Bantwal K, Wadhe V, Kulkarni A, Kulkarni S, Rajan MGR. A Study of Microalbuminuria (MAU) and Advanced Glycation End Products (AGEs) Levels in Diabetic and Hypertensive Subjects. Indian J Clin Biochem. 2018 Jan;33(1):81-85. doi: 10.1007/s12291-017-0638-5. Epub 2017 Feb 1. PMID 29371774
- [Background] Adamska E, Kretowski A, Goscik J, Citko A, Bauer W, Waszczeniuk M, Maliszewska K, Paczkowska-Abdulsalam M, Niemira M, Szczerbinski L, Ciborowski M, Gorska M. The type 2 diabetes susceptibility TCF7L2 gene variants affect postprandial glucose and fat utilization in non-diabetic subjects. Diabetes Metab. 2018 Sep;44(4):379-382. doi: 10.1016/j.diabet.2017.05.001. Epub 2017 May 31. No abstract available. PMID 28579156